CLINICAL TRIAL: NCT06436599
Title: Comparison of Serratus Posterior Superior Intercostal Plane Block Versus Deep Serratus Anterior Plane Block for Postoperative Analgesia After Breast Surgery: a Prospective Randomized Study
Brief Title: SPSIPB Versus Deep SAPB for Analgesia After Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Burgac (Other)
Responsible Party: Sponsor-Investigator, Mustafa Burgac, principal investigator, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/0870
Record Dates: First submitted 2024-05-22; First posted 2024-05-31 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: single blind
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with serratus posterior superior intercostal plan block (Active Comparator): Serratus posterior superior intercostal plane block was applied to a certain group of patients for postoperative analgesia
  Interventions: Other: plane block with %0.25 30 ml bupivacaine
- Patients with serratus anterior plan block (Active Comparator): Serratus anterior plane block was applied to a certain group of patients for postoperative analgesia
  Interventions: Other: plane block with %0.25 30 ml bupivacaine

INTERVENTIONS:
Other: plane block with %0.25 30 ml bupivacaine — evaluation of the efficacy of two different plan blocks for postoperative analgesia
  Other Names: postoperative analgesia

SUMMARY:
The application of regional anaesthetic procedures in breast surgery is associated with a lower incidence of chronic pain, reduced morbidity, shorter hospital stay and less opioid requirement. Therefore, we aimed to compared the postoperative analgesic efficacy of Serratus Anterior Plan Block and Serratus Posterior Superior Intercostal Plan Block in breast surgery.

DETAILED DESCRIPTION:
Breast surgery is one of the most common operations performed by General Surgery and may be associated with acute postoperative pain. Acute postoperative pain is an independent risk factor for the development of chronic pain after mastectomy. Various regional anaesthetic procedures have been tried to achieve better acute pain control and thus less chronic pain. The use of regional anaesthetic procedures in breast surgery is associated with a lower incidence of chronic pain, reduced morbidity, shorter hospital stay and less opioid requirement.

Interfascial plane blocks have become popular because they are easy to perform and safe. Since interfascial plan blocks are based on the injection of local anaesthetic between two fasciae, the complication rate such as nerve damage is very low. With this method, effective analgesia can be provided in various areas such as abdominal, thoracic and lumbar regions while reducing opioid consumption and avoiding neuraxial methods.

In randomised controlled trials investigating the efficacy of Serratus Anterior Plane Block for postoperative analgesia management after breast surgery, adequate analgesia was reported.

Serratus posterior superior intercostal plan block, a newly defined interfascial plan block, has been shown to provide a wide sensory blockade between intercostal muscles. Postoperative analgesic efficacy has been demonstrated in thoracic, breast and shoulder surgeries.

The aim of our study was to compared the postoperative analgesic efficacy of Serratus Anterior Plan Block and Serratus Posterior Superior Intercostal Plan Block in breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* unilateral mastectomy(modified radial mastectomy)
* ASA I-III risk group

Exclusion Criteria:

* Coagulopathy
* Wound and infection in the block area
* Local anaesthetic allergy
* Mental retardation
* Non-cooperative
* Pregnant patients

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of analgesic efficacy of postoperative plan blocks with numerical pain score (NRS) | within 24 hours postoperative
  Evaluation of which of the two plan blocks is more effective in postoperative analgesia.
  Postoperative pain scores will be evaluated with a numerical pain score. Evaluation will be performed postoperatively at 30. minutes, 1. hour, 4. hours, 8. hours, 12. hours and 24. hours. A lower numeric pain scale indicates a lower level of pain.

SECONDARY OUTCOMES:
Comparison of tramadol(mg) consumption | within 24 hours postoperative
  Using a patient-controlled analgesia device, tramadol consumption and total tramadol consumption will be compared between 0-1st hour, 1st-4th hour, 4th-8th hour, 8th-12th hour, 12th-24th hour postoperatively..
perioperative remifentanil consumption | perioperative
  The amounts (mcg) of remifantanil consumed during the surgical procedure will be compared
rescue anesthesia | within 24 hours postoperative
  In the postoperative 24-hour period, tenoxicam will be administered and recorded as rescue analgesia to patients who feel pain despite patient-controlled nalgesia (tramadol).
postoperative nausea-vomiting (PONV) | within 24 hours postoperative
  The number of times of nausea and vomiting in the postoperative period will be recorded and compared in both patient groups. A lower numerical value of postoperative nausea-vomiting indicates better patient comfort in the postoperative period.
surgeon and patient satisfaction (5-point Likert scale) | 24 hours after surgery
  At postoperative discharge, 5-point Likert satisfaction questionnaire will be administered to the surgeon and the patient. A high numerical value on a five-point Likert satisfaction scale indicates that the surgeon and the patient are satisfied with the procedure performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Professor Doctor Süleyman Yalçın City Hospital, Istanbul, Turkey (Türkiye)